CLINICAL TRIAL: NCT07282392
Title: Evaluating the Feasibility and Efficacy of Emotional Awareness and Expression Therapy (EAET) on Fibromyalgia Outcomes in Patients With Systemic Lupus Erythematosus (SLE).
Brief Title: Helping Lupus Patients Manage Fibromyalgia Symptoms Through Emotional Awareness and Expression Therapy (EAET)
Acronym: EAET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Dan Kaufmann, Ph.D., Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00194480
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lupus; Fibromyalgia (FM); Chronic Widespread Pain
Keywords: lupus; fibromyalgia; chronic widespread pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Awareness and Expression Therapy (Experimental): The treatment will be conducted via HIPAA-compliant video telemedicine (Zoom) in small groups of patients for eight weekly sessions, 2 hours per session. Each session will use an educational lecture, discussion, in-class experiential exercises, and homework assignments. During sessions, participants will be encouraged to identify their stressors and experiences, and to express their avoided or suppressed emotions, using exercises such as emotional disclosure, role-playing, and the "empty chair" technique. Participants will be given homework assignments to complete between sessions, including expressive writing, identifying stressors and avoided emotions, and practicing healthy communication skills.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy (EAET)
- Wait list control (No Intervention): Participants assigned to the waitlist control condition will be assessed at baseline and at a time matched to EAET post-treatment. All interested participants will be offered the opportunity to receive the EAET treatment once their WL period is completed. Those who opt to receive the treatment will be required to complete another set of assessments post-treatment.

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy (EAET) — EAET is a novel psychotherapy based on the well-supported finding that adverse, stressful, or traumatic life experiences result in maladaptive emotional experiences that can trigger or amplify pain and other symptoms. EAET showed promising results in fibromyalgia and migraines, as well as musculoskeletal pain, and was found to be more efficacious than CBT, the recommended treatment for chronic pain.
  Arms: Emotional Awareness and Expression Therapy

SUMMARY:
The goal of this clinical trial is to learn if a psychotherapy intervention works to relieve widespread pain in patients with lupus. The main questions it aims to answer are:

Is the psychotherapy treatment safe for lupus patients? Are lupus patients able to complete the treatment? Can the treatment help improve chronic pain and other symptoms in lupus patients?

Researchers will compare the treatment to a control (participants who will continue their medical treatment but will not receive psychotherapy for the time frame of the treatment) to see if the psychotherapy treatment works to relieve widespread pain and other lupus-related symptoms.

Participants will:

Fill out questionnaires before and after the treatment. Participate in 8 weekly treatment sessions, 2 hours per session, delivered via Zoom from their own home.

Keep a list of medications and monitor any changes in their medication regimen.

DETAILED DESCRIPTION:
Lupus is a serious and lifelong illness, causing flare-ups and damage to organs. It leads to a higher risk of death and a lower quality of life. Difficult life experiences, such as trauma or childhood adversity, are more common in people with lupus and fibromyalgia. These early experiences also raise the risk of anxiety, depression, and developing lupus later in life.

This study will test a new therapy, Emotional Awareness and Expression Therapy (EAET). EAET helps people understand and express emotions related to difficult past experiences, which may reduce physical pain and improve overall health. This study wants to see if EAET will help people with lupus who also suffer from chronic widespread pain (or fibromyalgia) and is safe.

Participants in the study will be randomly assigned to receive EAET therapy via telehealth or to a waiting list. The study will see if the treatment helps reduce lupus flares, pain, fatigue, anxiety, depression, and improve quality of life and sleep. The EAET group will attend eight two-hour online group therapy sessions once a week for 8 weeks. This group will also complete homework for about 30 minutes a day during participation. The wait list group will wait for 8 weeks until the EAET group is done. Both groups will complete surveys. The wait list group can choose to participate in the next therapy group session.

ELIGIBILITY:
Inclusion Criteria:

* Adults of all genders, ages 18-65.
* A diagnosis of lupus and fibromyalgia or chronic widespread pain by a licensed rheumatologist
* Be on a stable medication regimen.

Exclusion Criteria:

* Serious psychiatric disorders (e.g., schizophrenia or bipolar disorder) uncontrolled with medications.
* Active suicidal ideation.
* Untreated alcohol or substance use disorder.
* Substantial cognitive impairment.
* Changes in medications in the past 3 months.
* Enrollment in another treatment study.
* Current involvement in health-related litigation or disability application.
* Inability to use a computer and/or smartphone.
* limited access to the internet.
* Inability to communicate in English.
* Failure to complete the baseline assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2028-11-04 (Estimated)

PRIMARY OUTCOMES:
Widespread pain index at baseline | From enrollment to the end of treatment at 8 weeks
  A licensed rheumatologist will ask participants to identify 19 areas where they felt pain over the past week. The score ranges from 0 to 19 (the number of bodily regions).
Widespread pain index a week after treatment compared to baseline | 9 weeks after commencement of treatment
  A licensed rheumatologist will ask participants how many body areas they felt pain in during the week after treatment. The score ranges from 0 to 19, and the change in score will be compared with the baseline score. A lower score after treatment indicates the treatment's effectiveness in reducing widespread pain.
Symptom Severity Score at baseline | 1 week before the treatment
  A licensed rheumatologist will evaluate the symptom severity and somatic symptoms over the past week at baseline using a 0-3 scale.
Change in the severity scale after treatment compared to baseline. | 9 weeks after commencement of treatment
  A change in symptom severity will be evalauted by comparing the symptom severity score after treatment to baseline. A lower severity score after treatment indicates the treatment's effectiveness in reducing somatic symptoms.

SECONDARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) at baseline. | A week before treatment
  A licensed rheumatologist will evaluate the disease activity using the SLEDAI questionnaire at baseline. The scale ranges from 0 to 105. 0 indicates no disease activity; 1-5, mild disease activity; 6-10, a clinically meaningful cutoff indicating moderate disease activity; 11-19, high disease activity; and 20 or more, very high disease activity.
Change in SLEDAI measure after treatment compared to baseline. | 9 weeks after commencement of treatment
  A licensed rheumatologist will evaluate the disease activity using the SLEDAI questionnaire after treatment. A lower score after treatment indicates the treatment's effectiveness in reducing lupus disease activity.
Lupus-specific quality of life (LupusQol) index at baseline. | 1 week before commencement of treatment
  Lupus-related quality of life will be evaluated using the LupusQol questionnaire, which participants will complete. Scores range from 0 to 100. Higher scores indicate a higher quality of life.
Change in lupus-related quality of life after treatment compared to baseline. | 9 weeks following commencement of treatment
  Changes in Lupus-related quality of life will be evaluated by comparing scores on the LupusQol questionnaire after treatment with baseline scores. Higher scores indicate that the therapy increased participants' quality of life.
Fatigue at baseline | 1 week before commencement of treatment
  Fatigue will be evaluated at baseline using the patient-administered Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue). The score ranges from 0 to 52. A higher score indicates higher fatigue.
Change in fatigue score after treatment compared to baseline. | 9 weeks following commencement of treatment
  The FACIT-Fatigue scale will be administered after treatment, and the score will be compared with the baseline. A lower score indicates that the therapy improved fatigue.
Anxiety levels at baseline. | 1 week before the treatment.
  Anxiety will be measured using the Patient Reported Outcome Measurement Information System (PROMIS) short anxiety questionnaire. The minimum value is 8, and the maximum value is 40. A higher score on this test indicates higher levels of anxiety.
Change in anxiety levels after treatment compared to baseline. | 9 weeks after commencement of treatment
  A change in anxiety will be evaluated by comparing the PROMIS anxiety questionnaire score after treatment to baseline. A lower anxiety score after treatment will indicate the effectiveness of treatment in reducing anxiety.
Depression levels at baseline. | 1 week before treatment
  Depression will be measured using the Patient Reported Outcome Measurement Information System (PROMIS) short depression questionnaire. The minimum score is 8, and the maximum score is 40. A higher score indicates a higher level of depression.
Change in depression after treatment compared to baseline. | 9 weeks after commencement of treatment.
  A Change in depression score will be evaluated by comparing the PROMIS depression questionnaire score after treatment vs. baseline. A lower score will indicate the effectiveness of treatment in relieving depression.
Sleep disturbance at baseline. | 1 week prior to the commencement of therapy
  Sleep disturbance will be evalauted using the patient-administered PROMIS- sleep disturbance short form. The scores range from 8 to 40, with higher scores indicating a greater severity of sleep disturbance.
Change in sleep disturbance after treatment compared to baseline. | 9 weeks after the commencement of treatment
  The sleep disturbance score will be collected after treatment and compared with the baseline score. A lower score indicates that the therapy reduced sleep disturbance.
Sleep-related impairment at baseline. | 1 week before commencement of treatment
  Sleep-related impairment will be evalauted using the participant-administered PROMIS sleep-related impairment short form 8a. The scores range from 8 to 40, with higher scores indicating greater sleep-related impairment.
Change in sleep impairment after treatment compared to baseline. | 9 weeks after commencement of treatment.
  Sleep-related impairment will be scored after treatment and compared to the baseline score. A reduction in overall score indicates that the treatment was effective in reducing sleep-related impairment.

OTHER OUTCOMES:
Satisfaction with therapy and therapist. | 8 weeks after commencement of treatment
  Satisfaction with therapy and the therapist will be evaluated using the STTS-R inventory. Scores range from 13 to 65. Higher scores indicate higher satisfaction with therapists and treatment.
Satisfaction from the telemedicine questionnaire. | 8 weeks after commencement of treatment.
  Participants will complete the Satisfaction with telemedicine questionnaire, which assesses participants' satisfaction with the telehealth platform. The scores range from 14 to 70, with higher scores indicating greater satisfaction with telehealth.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Kaufmann, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yarns BC, Jackson NJ, Alas A, Melrose RJ, Lumley MA, Sultzer DL. Emotional Awareness and Expression Therapy vs Cognitive Behavioral Therapy for Chronic Pain in Older Veterans: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2415842. doi: 10.1001/jamanetworkopen.2024.15842. PMID 38869899
- [Background] Yarns BC, Lumley MA, Cassidy JT, Steers WN, Osato S, Schubiner H, Sultzer DL. Emotional Awareness and Expression Therapy Achieves Greater Pain Reduction than Cognitive Behavioral Therapy in Older Adults with Chronic Musculoskeletal Pain: A Preliminary Randomized Comparison Trial. Pain Med. 2020 Nov 1;21(11):2811-2822. doi: 10.1093/pm/pnaa145. PMID 32451528
- [Background] Lumley MA, Schubiner H, Lockhart NA, Kidwell KM, Harte SE, Clauw DJ, Williams DA. Emotional awareness and expression therapy, cognitive behavioral therapy, and education for fibromyalgia: a cluster-randomized controlled trial. Pain. 2017 Dec;158(12):2354-2363. doi: 10.1097/j.pain.0000000000001036. PMID 28796118